CLINICAL TRIAL: NCT06342635
Title: Prospective Observational Single-centre Study on the Efficacy and Safety of Hydra Transcatheter Aortic Valve
Brief Title: Hydra Single-centre Experience - Copenhagen, Denmark
Status: Recruiting | Type: Observational
Sponsor: Sahajanand Medical Technologies Limited (Industry)
Collaborators: Qmed Consulting A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: HYD/DENMARK-001/2023
Record Dates: First submitted 2024-03-21; First posted 2024-04-02 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Aortic Valve Stenosis
Keywords: Aortic Valve Stenosis; TAVI; Hydra
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Hydra Transcatheter Aortic Valve (THV) Series — The Hydra device consists of a self-expanding nitinol frame and three bovine pericardial leaflets in supra-annular position.

SUMMARY:
The present study aims to evaluate the efficacy and safety of TAVI using the Hydra transcatheter aortic valve (THV) series, in patients with severe aortic stenosis up to 1-year after the procedure. Additionally, the study will assess the role of geometry in the development of new conduction abnormalities based on the analysis of post-operative CT scan at 1-month in patients who had undergone transcatheter aortic valve replacement with a self-expanding Hydra THV series.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patients affected by severe aortic stenosis (NYHA class ≥ II) eligible for TAVI procedure as per local Heart Team evaluation
3. Full understanding and willing to provide informed consent to study enrolment

Exclusion Criteria:

1. Contraindications to TAVI (e.g., anatomically phenotypes, intracardiac mass, thrombus, vegetation, endocarditis)
2. Refusal to provide informed consent to study enrolment
3. Patients with severe aorta or peripheral artery disease precluding transfemoral approach of TAVI
4. Patients with calcification on the annulus and in the Left Ventricular Outflow Tract (LVOT), or/and excess calcium within each cusp, or those who are deemed unsuitable for the Hydra THV series based on the clinical judgment of the Investigator

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with severe aortic valve stenosis
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Primary safety endpoint | 30 days
  Early safety as defined by VARC-3, as composite of:
  * Freedom from all-cause mortality;
  * Freedom from all stroke;
  * Freedom from VARC 3 type 3-4 bleeding;
  * Freedom from major vascular, access-related, or cardiac structural complication;
  * Freedom from acute kidney injury stage 3 or 4;
  * Freedom from moderate or severe aortic regurgitation;
  * Freedom from new permanent pacemaker due to procedure-related conduction abnormalities;
  * Freedom from surgery or intervention related to the device.
Primary performance endpoint | 30 days
  Device success as defined by VARC-3, as composite of:
  * Technical success;
  * Freedom from mortality;
  * Freedom from surgery or intervention related to the device or to a major vascular or access related or cardiac structural complication;
  * Intended performance of the valve (mean gradient <20mmHg, peak velocity <3 m/s, Doppler velocity index ≥0.25, and less than moderate aortic regurgitation).

SECONDARY OUTCOMES:
Technical success | Immediately after procedure
Cardiovascular mortality | 30 days, and 1-year
All-cause mortality | 30 days, and 1-year
All stroke | 30 days, and 1-year
Disabling stroke | 30 days, and 1-year
Myocardial infarction | 30 days, and 1-year
Major vascular complication | 30 days
Acute kidney injury | 30 days
New permanent pacemaker implantation due to procedure related conduction abnormalities | 30 days, and 1-year
New-onset atrial fibrillation | 30 days, and 1-year
Coronary artery obstruction requiring intervention | 30 days, and 1-year
Re-hospitalization for procedure- or valve-related causes | 30 days, and 1-year
Mean aortic valve gradient | 30 days, and 1-year
Effective Orifice Area (EOA) | 30 days, and 1-year
Paravalvular leak | 30 days, and 1-year
New York Heart Association (NYHA) functional class | 30 days, and 1-year
Quality-of-life evaluation | 30 days, and 1-year
Bioprosthetic Valve Failure (BVF) | 30 days, and 1-year
Bioprosthetic valve dysfunction (BVD) | 30 days, and 1-year
Stroke or peripheral embolism | 30 days, and 1-year
VARC-3 Type 3-4 bleeding secondary to or exacerbated by antiplatelet or anticoagulant agents used specifically for valve-related concerns | 30 days, and 1-year
Rates of Hypoattenuated Leaflet Thickening (HALT) | 30 days
Rates of Reduced leaflet motion (RLM) | 30 days
Commissural alignment | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark